CLINICAL TRIAL: NCT02316158
Title: PsYoungSupport Internet and Communication Technology Based Health Programmes - Information, Education and Support to Young People Close to Persons With Mental Illness
Brief Title: PsYoungSupport - Web-based Support to Young Careers to Persons With Mental Illness
Acronym: PSYS
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Vardalinstitutet The Swedish Institute for Health Sciences (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: A2007003
Record Dates: First submitted 2011-09-02; First posted 2014-12-12 (Estimated); Last update posted 2014-12-12 (Estimated); Status verified 2011-09

CONDITIONS: Mental Illness; Web
Keywords: Burden; Mental illness; Stress; Social support
MeSH Terms: conditions — Mental Disorders

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Webb-based support and education (Experimental): It contains of two parts 1) evidence based information (about mental diseases, early signs, coping strategies, what you can do for your relative or close friend, what you can do for yourself, addresses to networks and web sites, relevant juridical issues, etc), 2) FAQ, where you directly can find answers to common questions.
  Interventions: Other: Web-based support
- Available support in society (Active Comparator): Available support in society for young persons presented in a brochure
  Interventions: Other: Web-based support

INTERVENTIONS:
Other: Web-based support — Comparison between the efficacy between webb-based support and informational support
  Other Names: website: www.molnhopp.nu

SUMMARY:
The overall aim with the project PsYoungSupport is to evaluate Internet and communication technology (ICT) health efforts, i.e. information, education and support for young adults (16-25 years) who are first degree relatives or represent the close social network (relative or close friend) of individuals with mental illness, with regard to the process (the quality and usefulness of the support) and the effect (on health and quality of life, situation as relative or part of close social network and consumption of other support/care) of the intervention.

The participatory design is one of the foundations of this project, and young adult participants will be consulted through out the research project. PsYoungSupport is a research program comprising three phases, Phase I is a survey of young relatives' and close friends' needs for internet based information, education and support, Phase II is the development of a website, and Phase III is an intervention based on the previous phases. The aim of phase III is to evaluate the effect of an internet based intervention containing information, education and support for young adults in families where a family member suffers from mental illness or functional disability. The participants (N=400) will be randomised to two groups with different kinds of support. The participants will be evaluated using self-questionnaires and web interviews at the following occasions: baseline at the start of the intervention, after 4 months and after 8 months. This project will have implications for persons suffering from mental illness as well as for their relatives and close friends.

DETAILED DESCRIPTION:
In the last decades it has been stated that the mental health of young people has deteriorated. Nowadays, the main part of the psychiatric care are out-patient care, family, relatives and close friends get involved and needs to take large responsibility for their relative or friend with mental illness. Therefore it is important to acquire knowledge that could benefit the patients and their families. There is still a gap in the knowledge as to which social support, such as information and education processes, are of value to the patient and family struggling with depression, and as to how individuals benefits from these components in their functional recovery from depression. Accordingly, pedagogic processes as an integrated part of patient-centred care and treatment may be increasingly important to study.

The overall aim is to evaluate internet and communication technology (ICT) health efforts, i.e. information, education and support for young adults who are first degree relatives or represent the close social network (relative or close friend) of individuals with mental illness, with regard to the process (the quality and usefulness of the support) and the effect (on health and quality of life, situation as relative or part of close social network and consumption of other support/care) of the intervention.

PsYoungSupport is a research program comprising three phases, Phase I is a survey of young relatives' and close friends' needs for internet based information, education and support, Phase II is the development of a website, and Phase III is an intervention based on the previous phases. The investigators have a participatory design, including young persons in the whole research process. Primary outcome measures are social interaction, the degree of subjective and objective burden, stigmatisation and illness. Data are going to be based on both qualitative and quantitative approaches. The results are also going to evaluate cost effectiveness and the process of learning.

Within three years this project will describe different kind of implications for relatives and close friends who are caring for persons suffering from mental illness. Increased accessibility to knowledge about how mental health can benefit them and their relatives and close friends will facilitate for and empower these persons, and also increase their participation in society and with that increase the democracy for these persons in the society. Within five years this study can be integrated within the Swedish national website Care on line.

ELIGIBILITY:
Inclusion Criteria:

* age 16-25 years
* seeing themselves as a relative or close friend who supports a person with mental illness

Exclusion Criteria:

* persons who do not understand, read or express him-/herself in Swedish
* persons with acute severe mental illness or acute suicidal risk

Ages: 16 Years to 25 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 241 (Actual)
Dates: Start 2009-03; Primary Completion 2009-06 (Actual); Study Completion 2010-05 (Actual)

PRIMARY OUTCOMES:
Decreased change in Burden | 8 months
  Cope Index (McKee, Philp, Lamura et al 2003. The Cope Index measures components such as negative effect of caring, positive values and the quality of support aspects of supporting a relative or close friend. Each question is answered on a 4-point scale with the alternative 'never' ,'sometimes', 'often' and 'always'. Some questions have the alternative of 'not applicable'. All scores are added within each area and high scores indicate a high level of negative effect, positive value and quality of support.

SECONDARY OUTCOMES:
Decreased Stress | Eight months
  Perceived Stress Scale (Cohen Kamch, Meremelstein, 1983). Measures the degree to which situations in individuals' daily life are appraised as stressful. The questions cover how the informant felt and thought during the last month. The questionaire consist of 10 items and each item is answered on a 5-point scale 0=never; 1=almost never; 2=sometimes; 3=faily often and 5=very often. PSS scores are obtained by reversing responses (e.g., 0=4; 1=3; 2=2; 3=1 and 4=0 to the 4 positively stated items (items 4,5,7 & 8) and then summing across all scale items

CONTACTS AND LOCATIONS:
Overall Officials: Ingela Skärsäter, PhD, Principal Investigator — University of Gothenburg, 405 30 Göteborg, Sweden; Barbro Krevers, PhD, Principal Investigator — Linköping University, 581 83 Linköping, Sweden
Locations (1):
- Vårdalinstitutet - The Swedish Institute for Health Sciences, Gothenburg, Sweden